CLINICAL TRIAL: NCT02379104
Title: ROTEM® Sigma Performance Evaluation - Method Comparison With Predicate Device and Reference Intervals
Acronym: ROSI-EVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tem Innovations GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RSE2015
Record Dates: First submitted 2015-02-12; First posted 2015-03-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Blood Coagulation Disorders
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers fulfilling inclusion/exclusion criteria for reference interval sample group are tested with ROTEM sigma
  Interventions: Device: ROTEM sigma
- Patients with expected coagulopathy: Patients with expected bleeding and coagulation problems during elective surgery or at the ICU, or trauma patients are tested with ROTEM sigma and ROTEM delta comparatively
  Interventions: Device: ROTEM sigma

INTERVENTIONS:
Device: ROTEM sigma — Group Healthy Volunteers: a blood sample is tested with ROTEM sigma Group Patients with expected coagulopathy: a blood sample is tested with ROTEM sigma and ROTEM delta in parallel
  Other Names: ROTEM delta

SUMMARY:
ROTEM® sigma is a new thromboelastometric coagulation analysis system. The new system is fully automated allowing for a simple and safe operation compared to its predecessor model ROTEM® delta.

Method comparison of ROTEM® sigma with predecessor model ROTEM® delta) - confirmation of equality.

Confirmation of reference intervals of the ROTEM® systems.

DETAILED DESCRIPTION:
The main innovation of ROTEM® sigma is the development of a sample handler and a cartridge allowing for a of full automated test operation. As in ROTEM® delta four different tests can be run simultaneously on the four channels of the analyser.

Whereas the tests in ROTEM® delta are performed manually by pipetting a blood sample and liquid system reagents, in ROTEM® sigma the reagents are contained in freeze dried pellet form in a cartridge. Test operation is performed by inserting a cartridge and attaching a blood sample to the analyser.

The five available ROTEM® tests INTEM, EXTEM, FIBTEM, APTEM, and HEPTEM are contained in different combinations in two cartridge configurations:

* Cartridge type 1 including INTEM, EXTEM, FIBTEM, APTEM
* Cartridge type 2 including INTEM, EXTEM, FIBTEM, HEPTEM

Aim of the study is the performance evaluation of the new ROTEM® sigma coagulation analyzer in comparison to the current ROTEM® delta thromboelastometry system.

As a valid method comparison requires test results that cover the whole measurement range of the test system it is also necessary to include acute bleeding and emergency patients in the study. Only the inclusion of acute bleeding and emergency patients will produce strong pathologic test results allowing for a valid evaluation of the test system.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age ≥ 18 years
* Informed written consent
* Patients with an acute bleeding during surgery
* Or: trauma patients with acute bleeding
* Or: hypercoagulable (above normal fibrinogen) patients at the ICU

Healthy Volunteers:

* Adult healthy individuals (≥ 18 years)
* Written informed consent

Exclusion Criteria:

Patients:

• none

Healthy Volunteers:

* Any indications of alcohol or illegal drug abuse
* Any chronic disease with possible effect on the coagulation (liver disease, coronary heart disease)
* Any acute illness within the last 14 days
* Any hemostasis associated disease (myocardial infarction, thrombosis , stroke etc.) within the last year
* Intake of any coagulation affecting medication (aspirin, pain-killers, anti-rheumatic drugs, marcumar, platelet inhibitors) within the last 14 days
* Females only: known pregnancy
* Females only: breast feeding
* Any indication for any hemostasis disorder as interrogated by a specific history of bleeding tendencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with expected bleeding and coagulation problems during elective surgery or at the ICU, or trauma patients
  * Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Method comparison: linear regression analysis and bias estimation at medical decision limits | Parameter differences assessed at time of blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Volker Friemert, Dr., Study Chair — Tem Innovations GmbH
Locations (5):
- United States (3):
  - Florida Hospital Center for Thrombosis Research, Orlando, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Department of Anesthesiology Weill Cornell Medical College New York-Presbyterian Hospital, New York, New York
- Medi. Medical University Innsbruck Department of General and Surgical Intensive Care Medicine, Medical University Innsbruck, Innsbruck, Austria
- Institute of Anaesthesiology, Section Anaesthesiology, Intensive Care Medicine and OR-Management University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No